CLINICAL TRIAL: NCT00004158
Title: A Phase I/II Study of Targeted Radiotherapy Using Holmium-166-DOTMP With Melphalan and Peripheral Blood Stem Cell Transplantation for Treatment of Multiple Myeloma
Brief Title: Radiation Therapy Using Holmium Ho 166 DOTMP Plus Melphalan and Peripheral Stem Cell Transplantation in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1442.00; FHCRC-1442.00; NEORX-9804; NCI-G99-1623; CDR0000067396 (Registry Identifier: PDQ)
Record Dates: First submitted 1999-12-10; First posted 2004-07-19 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Melphalan; Peripheral Blood Stem Cell Transplantation; holmium-1,4,7,10-tetraazacyclododecane-N,N',N'',N'''-tetrakis(methylenephosphonic acid)

INTERVENTIONS:
Drug: melphalan
Procedure: peripheral blood stem cell transplantation
Radiation: holmium Ho 166 DOTMP

SUMMARY:
RATIONALE: Radiation therapy using holmium Ho 166 DOTMP may damage cancer cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy used to kill cancer cells.

PURPOSE: Phase I/II trial to study the effectiveness of radiation therapy using holmium Ho 166 DOTMP plus melphalan and peripheral stem cell transplantation in treating patients who have multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of targeted radiotherapy using holmium Ho 166 DOTMP when combined with melphalan and autologous or syngeneic peripheral blood stem cell transplantation in patients with multiple myeloma. II. Determine the response rate and time to progression in patients treated with this regimen.

OUTLINE: This is a dose escalation, multicenter study of targeted radiotherapy using holmium Ho 166 DOTMP. Phase I: Autologous or syngeneic peripheral blood stem cells (PBSC) are harvested and selected for CD34+ cells. Patients receive an initial test dose of holmium Ho 166 DOTMP IV. Patients with adequate skeletal uptake of the test dose then receive therapeutic dose holmium Ho 166 DOTMP IV over 5-10 minutes for 1-3 days beginning 2 days after test dose infusion and melphalan IV over 20-30 minutes on day -3. PBSC are reinfused beginning a minimum of 24 hours after melphalan infusion and after ongoing radiation to bone marrow falls to less than 1 rad/hour. Cohorts of 4-7 patients receive escalating doses of targeted radiotherapy using holmium Ho 166 DOTMP until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 7 patients experience dose limiting toxicity. Phase II: Patients receive holmium Ho 166 DOTMP at the MTD from phase I of the study. Patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Multiple myeloma with one of the following: Complete or partial response to initial chemotherapy OR Primary refractory disease OR Chemotherapy responsive relapse Undergoing autologous or syngeneic peripheral blood stem cell transplantation No myeloma in refractory relapse

PATIENT CHARACTERISTICS: Age: 18 to physiologic 65 Performance status: Zubrod 0-2 Life expectancy: Not severely limited by concurrent illness Hematopoietic: Not specified Hepatic: Bilirubin less than 2 mg/dL SGPT less than 4 times normal Renal: Creatinine clearance at least 30 mL/min Cardiovascular: No uncontrolled arrhythmias or symptomatic cardiac disease Pulmonary: No symptomatic pulmonary disease FEV1, FVC, and DLCO at least 50% of predicted Other: Not pregnant or nursing Fertile patients must use effective contraception HIV negative No spinal cord compression

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Prior external beam radiotherapy not to exceed 30 Gy to spinal cord or greater than 20% of bone marrow volume Surgery: Not specified Other: At least 1 month since prior bisphosphonates No other concurrent experimental agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-06; Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William I. Bensinger, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (4):
- United States (4):
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington